CLINICAL TRIAL: NCT06527638
Title: PURI-PRO (Portuguese URinary Incontinence PROject) - Symptoms Impact and eHealth Intervention for Menopausal Women With Urinary Incontinence
Brief Title: PURI-PRO - Symptoms Impact and eHealth Intervention for Menopausal Women With Urinary Incontinence
Acronym: PURI-PRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Marta Monteiro da Silva Gonçalves Porto, Principal Investigator, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D-022-11-2019
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Menopause; Quality of life; Sexual Function; Beliefs and Coping Strategies; Social Isolation; Self Esteem; Pelvic Floor Muscle Training
MeSH Terms: conditions — Urinary Incontinence; Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth intervention for UI symptoms improvement (Experimental): Participants in the Experimental Group were integrated into an eHealth 8-week group intervention, based on the Health Action Process Approach (HAPA).
  The eHealth (internet-based) cognitive-behavioural intervention developed to promote UI symptoms improvement consisted of: i) weekly group sessions (by Zoom platform), with a specific theme in each session, ii) weekly challenges, and iii) WhatsApp group interaction.
  Interventions: Behavioral: Experimental Group: eHealth intervention for UI symptoms improvement
- Control Group: Delivery of a Health Literacy single-leaflet (Active Comparator): The control group received a health literacy single-leaflet, delivered through email.
  Interventions: Behavioral: Control Group: Delivery of a Health Literacy single-leaflet

INTERVENTIONS:
Behavioral: Experimental Group: eHealth intervention for UI symptoms improvement — The intervention was theoretically based on the HAPA model (including effective strategies in behaviour change, for example, action planning and coping with obstacles) and Common Sense Model of Self Regulation (beliefs, coping and appraisal), focusing on risk perception, planning, and self-efficacy.
  The intervention consisted of 8 sessions (90 minutes, once a week). All group intervention sessions, through the Zoom platform, were led by the psychologist responsible for the study, except the second session that was led by a physiotherapist. WhatsApp groups were created, to share experiences, knowledge, doubts and fears, and to create a sense of belonging, understanding and cohesion.
  All primary and secondary outcome measures were assessed at baseline, mid-intervention (one month later), post-intervention, and in a 3 month follow-up after the intervention.
  Arms: eHealth intervention for UI symptoms improvement
Behavioral: Control Group: Delivery of a Health Literacy single-leaflet — A health literacy single-leaflet was delivered, by e-mail in the first week of the intervention. Beyond this, there was no further interaction with the group.
  All primary and secondary outcome measures were assessed at baseline, mid-intervention (one month later), post-intervention, and in a 3 month follow-up after the intervention.
  Arms: Control Group: Delivery of a Health Literacy single-leaflet

SUMMARY:
Urinary Incontinence (UI) is a public health problem that disrupts the Quality of Life, Productivity, Social Isolation and Sexual Function; its prevalence in peri- and postmenopausal women is around 30-40%. UI remains underreported and undertreated. Previous eHealth interventions have been efficacious with women.

Thus, PURI-PRO (Portuguese Urinary Incontinence Project) (FCT Grant 2020.05710.BD) entailed a low-cost 8-week eHealth cognitive-behavioural multidisciplinary intervention aimed at reducing UI symptoms' severity through Pelvic Floor Muscle Training, development of healthy bladder habits, and promotion of adherence to exercises, realistic UI-beliefs, and functional coping strategies.

Urinary incontinence symptom severity, frequency and its impact on quality of life, beliefs and strategies regarding urinary incontinence, self-esteem, social isolation, and adherence to pelvic floor muscle excercises were evaluated.

DETAILED DESCRIPTION:
PURI-PRO's intervention followed an experimental design (randomised controlled trial) involving UI intervention (Experimental Group-EG) vs. Health Literacy single-leaflet (Control Group-CG), both delivered through the internet (eHealth). The study was comparative, since the sample was distributed in two groups (EG vs CG) through randomised distribution, and longitudinal, since all the outcome measures were evaluated at four different times.

ELIGIBILITY:
Inclusion Criteria:

* Age (40-65 years);
* Sex (women);
* The presence of UI (positive response to a question about experiencing involuntary urine loss during intra-abdominal pressure increment and/or when feeling an incontrollable urge to urinate, occasionally or frequently);
* Internet access.

Exclusion Criteria:

* Pregnancy or delivery in the past 6 months;
* Previous UI-related surgery;
* History of pelvic prolapse:
* Known malignancy in the lower abdomen;
* Neurological disease that could affect bladder control;
* Substance use disorder.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Brief Assessment of Urinary Incontinence symptoms and impact of Quality of Life | Change from Baseline urinary incontinence symptoms and impact on quality of life adherence to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by "International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form" (ICIQ-UI SF)
UI-related Coping Strategies | Change from Baseline UI-related coping strategies to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by a bi-factorial instrument (hiding coping dimension and defensive coping dimension) developed by our team that entails a set of UI-related maladaptive coping strategies to manage immediate effects of UI. This instrument is based on the work of Diokno and collaborators.
UI-related Beliefs | Change from Baseline UI-related beliefs to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by the Portuguese version of the "Brief Illness Perception Questionnaire" (IPQ-Brief). This instrument is based on the work of Figueiras and collaborators.

SECONDARY OUTCOMES:
Urinary Incontinence symptom severity and impact | Change from Baseline Urinary Incontinence symptom severity and impact to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by "King´s Health Questionnaire" (KHQ)
Self-reported Quality of Life | Change from Baseline quality of life to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by the Portuguese version of the "WHO Quality-of-Life-Bref" (WHOQOL-Bref).
Behavior Change (HAPA) | Change from Baseline behavior to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by the HAPA Questionnaire (tailored to Urinary Incontinence symptoms), based on Renner's and Schwarzer's RACK study
Self-esteem | Change from Baseline self-esteem to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by the Rosenberg Self-Esteem Scale (RSS)
Social Isolation | Change from Baseline social isolation to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by "Social Isolation Questionnaire" (tailored to Urinary Incontinence symptoms) (UI-SIQ). This questionnaire is still on the process of being published by our team.
Pelvic Floor and UI Knowledge | Change from Baseline pelvic floor and UI knowledge to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by "Prolapse and Incontinence Knowledge Questionnaire" (PIKQ-UI)
Pelvic Floor Muscle Exercises Adherence | Change from Baseline pelvic floor muscle exercises adherence to mid-intervention (1 month later), post-intervention (2 months later), and at a 3 month follow-up
  Evaluated by a checklist developed by Alewijnse and collaborators that includes items regarding the frequency, ease and satisfaction towards the pelvic floor muscle exercises

CONTACTS AND LOCATIONS:
Overall Officials: Marta G Porto, Master's, Principal Investigator — ISPA-IU; Filipa F Pimenta, PhD, Study Chair — ISPA-IU
Locations (1):
- ISPA-IU, Lisbon, Portugal

REFERENCES:
- [Background] Schroe H, Van Dyck D, De Paepe A, Poppe L, Loh WW, Verloigne M, Loeys T, De Bourdeaudhuij I, Crombez G. Which behaviour change techniques are effective to promote physical activity and reduce sedentary behaviour in adults: a factorial randomized trial of an e- and m-health intervention. Int J Behav Nutr Phys Act. 2020 Oct 7;17(1):127. doi: 10.1186/s12966-020-01001-x. PMID 33028335
- [Background] Schwarzer R, Renner B. Social-cognitive predictors of health behavior: action self-efficacy and coping self-efficacy. Health Psychol. 2000 Sep;19(5):487-95. PMID 11007157
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Imamura M, Abrams P, Bain C, Buckley B, Cardozo L, Cody J, Cook J, Eustice S, Glazener C, Grant A, Hay-Smith J, Hislop J, Jenkinson D, Kilonzo M, Nabi G, N'Dow J, Pickard R, Ternent L, Wallace S, Wardle J, Zhu S, Vale L. Systematic review and economic modelling of the effectiveness and cost-effectiveness of non-surgical treatments for women with stress urinary incontinence. Health Technol Assess. 2010 Aug;14(40):1-188, iii-iv. doi: 10.3310/hta14400. PMID 20738930
- [Background] Harper RC, Sheppard S, Stewart C, Clark CJ. Exploring Adherence to Pelvic Floor Muscle Training in Women Using Mobile Apps: Scoping Review. JMIR Mhealth Uhealth. 2023 Nov 30;11:e45947. doi: 10.2196/45947. PMID 38032694
- [Background] Dumoulin C, Hay-Smith J, Frawley H, McClurg D, Alewijnse D, Bo K, Burgio K, Chen SY, Chiarelli P, Dean S, Hagen S, Herbert J, Mahfooza A, Mair F, Stark D, Van Kampen M; International Continence Society. 2014 consensus statement on improving pelvic floor muscle training adherence: International Continence Society 2011 State-of-the-Science Seminar. Neurourol Urodyn. 2015 Sep;34(7):600-5. doi: 10.1002/nau.22796. Epub 2015 May 21. PMID 25998603
- [Background] Garley A, Unwin J. A case series to pilot cognitive behaviour therapy for women with urinary incontinence. Br J Health Psychol. 2006 Sep;11(Pt 3):373-86. doi: 10.1348/135910705X53876. PMID 16870050
- [Background] Funada S, Watanabe N, Goto T, Negoro H, Akamatsu S, Ueno K, Uozumi R, Ichioka K, Segawa T, Akechi T, Furukawa TA, Ogawa O. Cognitive behavioral therapy for overactive bladder in women: study protocol for a randomized controlled trial. BMC Urol. 2020 Aug 20;20(1):129. doi: 10.1186/s12894-020-00697-0. PMID 32819331
- [Background] Steenstrup B, Lopes F, Cornu JN, Gilliaux M. Cognitive-behavioral therapy and urge urinary incontinence in women. A systematic review. Int Urogynecol J. 2022 May;33(5):1091-1101. doi: 10.1007/s00192-021-04989-3. Epub 2021 Oct 30. PMID 34716765
- [Background] Dowd T, Kolcaba K, Steiner R. Using cognitive strategies to enhance bladder control and comfort. Holist Nurs Pract. 2000 Jan;14(2):91-103. doi: 10.1097/00004650-200001000-00013. PMID 12119974
- [Background] Dumoulin C, Alewijnse D, Bo K, Hagen S, Stark D, Van Kampen M, Herbert J, Hay-Smith J, Frawley H, McClurg D, Dean S. Pelvic-Floor-Muscle Training Adherence: Tools, Measurements and Strategies-2011 ICS State-of-the-Science Seminar Research Paper II of IV. Neurourol Urodyn. 2015 Sep;34(7):615-21. doi: 10.1002/nau.22794. Epub 2015 May 21. PMID 25998493
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Bo K, Fernandes ACNL, Duarte TB, Brito LGO, Ferreira CHJ. Is pelvic floor muscle training effective for symptoms of overactive bladder in women? A systematic review. Physiotherapy. 2020 Mar;106:65-76. doi: 10.1016/j.physio.2019.08.011. Epub 2019 Aug 24. PMID 32026847
- [Background] Dowd T, Dowd ET. A cognitive therapy approach to promote continence. J Wound Ostomy Continence Nurs. 2006 Jan-Feb;33(1):63-8. doi: 10.1097/00152192-200601000-00010. PMID 16444107
- [Background] Kelleher CJ, Cardozo LD, Khullar V, Salvatore S. A new questionnaire to assess the quality of life of urinary incontinent women. Br J Obstet Gynaecol. 1997 Dec;104(12):1374-9. doi: 10.1111/j.1471-0528.1997.tb11006.x. PMID 9422015
- [Background] Alewijnse D, Metsemakers JF, Mesters IE, van den Borne B. Effectiveness of pelvic floor muscle exercise therapy supplemented with a health education program to promote long-term adherence among women with urinary incontinence. Neurourol Urodyn. 2003;22(4):284-95. doi: 10.1002/nau.10122. PMID 12808702
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Canavarro MC, Serra AV, Simoes MR, Rijo D, Pereira M, Gameiro S, Quartilho MJ, Quintais L, Carona C, Paredes T. Development and psychometric properties of the World Health Organization Quality of Life Assessment Instrument (WHOQOL-100) in Portugal. Int J Behav Med. 2009;16(2):116-24. doi: 10.1007/s12529-008-9024-2. Epub 2009 May 8. PMID 19424810
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Diokno AC, Burgio K, Fultz NH, Kinchen KS, Obenchain R, Bump RC. Medical and self-care practices reported by women with urinary incontinence. Am J Manag Care. 2004 Feb;10(2 Pt 1):69-78. PMID 15011807
- [Background] Shah AD, Massagli MP, Kohli N, Rajan SS, Braaten KP, Hoyte L. A reliable, valid instrument to assess patient knowledge about urinary incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1283-9. doi: 10.1007/s00192-008-0631-x. Epub 2008 May 15. PMID 18480958
- [Background] Figueiras, M. J., Monteiro, R., and Caeiro, R. (2012). Crenças erróneas e perceção da doença em pacientes cardíacos e seus cônjuges: Um estudo piloto. Psychol. Commun. Health 1, 232-245. https://doi.org/10.5964/pch.v1i3.24
- [Background] Renner B, Schwarzer R. Risk and health behaviors. Documentation of the scales of the research project: Risk appraisal consequences in Korea (RACK) 2nd ed. Bremen: International University Bremen & Freie Universität Berlin; 2005.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT06527638/ICF_000.pdf